CLINICAL TRIAL: NCT02636959
Title: High Volume Saline Irrigation in the Post-operative Management of Chronic Rhinosinusitis: A Multicenter Randomized Single-Blind Controlled Trial
Brief Title: A Postoperative Study on HVSI vs LVSI Treatment of Chronic Rhinosinusitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15-02550
Record Dates: First submitted 2015-12-02; First posted 2015-12-22 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- high volume saline irrigation (HVSI) (Active Comparator): High volume nasal spray, NeilMed® Sinus Rinse, is a high saline nasal rinse that is a safe, nonpharmacologic treatment. Randomized participants will be asked to use the rinse for one month (twice daily) by following the manufacturer's guidelines and use of the squeeze bottle provided. Preoperative and one month Postoperative sinus surgery, the participants will complete subjective questionnaires and at one-month after surgery, endoscopic sinonasal photos will be taken. These data will be used to assess the quality of postoperative improvements after treatment.
  Interventions: Other: saline irrigation
- low volume saline irrigation (LVSI) (Active Comparator): Low volume nasal spray, Salinex Rinse, is a low saline nasal rinse that is a safe, nonpharmacologic treatment. Randomized participants will be asked to use the rinse for one month (twice daily) by following the manufacturer's guidelines and use of the squeeze bottle provided. Preoperative and one month Postoperative sinus surgery, the participants will complete subjective questionnaires and at one-month after surgery, endoscopic sinonasal photos will be taken. These data will be used to assess the quality of postoperative improvements after treatment.
  Interventions: Other: saline irrigation

INTERVENTIONS:
Other: saline irrigation — HVSI (NeilMed® Sinus Rinse™) versus LVSI (Salinex®) in the early post-operative management in patients with chronic rhinosinusitis. Both are a saline rinse spray.

SUMMARY:
Chronic sinusitis (CRS) is a common inflammatory sinus condition among Canadians. Saline irrigation is an effective therapy used in the management of CRS and is a commonly prescribed treatment in preoperative surgery for people with this condition. Recently, a study performed by a Toronto group in Canada tried to show if there is any significant improvement between using high versus low volume saline irrigation to treat CRS. Despite finding a trend, the number of people with CRS used in this pilot study was not large enough to conclusively declare any difference between the two treatment groups.

PURPOSE: The purpose of this study is to determine if there is a clinical benefit of high volume saline nasal irrigation (HVSI) over low volume saline irrigation (LVSI) in the postoperative period in patients with chronic Rhinosinusitis (CRS). This study is part of a multicenter collaborative project initiated by Macdonald et al. (20). A sample size of 176 participants (88 in each condition) is required to achieve data significance. To achieve this, our role is to collect data (plus those of four other Canadian rhinology research centres) from 20 patients and add our findings to theirs to establish an acceptable and significant result. This information would help otolaryngologists, family physicians, and other health care professionals recommend the best post-operative SNI (saline nasal irrigation) device for their patients with CRS.

DETAILED DESCRIPTION:
BACKGROUND: Chronic Rhinosinusitis (CRS) is a common inflammatory condition of the upper respiratory tract lasting more than 8 to 12 weeks. Major symptoms include facial congestion/fullness, facial pain/pressure, nasal obstruction/blockage, purulent nasal drainage, and reduction or loss of smell. The diagnosis must include two major symptoms and either endoscopic evidence of polyps, edema or mucopurulent discharge from the middle meatus and/or CT changes in the mucosa of sinuses or osteomeatal complexes.

CRS has an estimated prevalence of 5% in the Canadian population, and up to 16% in some adult populations in the United States. Sinusitis is associated with a major societal health care burden, costing billions of dollars a year in North America. The medical treatment of CRS includes topical saline and corticosteroid sprays, systemic steroids and antimicrobials. Specifically, saline nasal irrigation (SNI) is a safe, nonpharmacologic treatment, and an important and efficacious component in the management of CRS. SNI can vary by concentration (e.g. hypertonic, isotonic, hypotonic) and device (e.g. bulb syringe, nasal mist, squeeze bottle).

The Mayo Clinic recently reviewed major expert consensus guidelines on the medical treatment of CRS. Although they recognized an overall paucity of controlled trials for any medical treatment, and a lack of a consensus or algorithm in the treatment of CRS, there is an overall consensus agreement of the use for SNI in this population. In this review, there was no mention of treatment of CRS in postoperative period, and no recommendation of what type of SNI is best.

Few studies examine various SNI formulations in the postoperative period. These were highlighted by Canadian authors in a recent exhaustive review of SNI in sinusitis. Three studies, all greater than 15 years old, include formulations that are not currently in popular use, or even available in North America. These did show that pressurized jets or sprays of seawater were more effective than nasal drops. More recently, Harvey et al. examined how irrigation is delivered and retained in the sinus, using more common devices. In a cadaveric model, they compared high volume saline nasal irrigation (HVSI) to low volume saline nasal irrigation (LVSI) devices and found a greater delivery (p<0.02) in the former. To date there are no studies comparing HVSI to LVSI, using subjective patient benefit and objective endoscopic measure outcomes, in the postoperative CRS patient.

One study did examine two different SNI devices in the management of CRS. The authors recruited 150 subjects with CRS in the primary care setting, and randomized them to two weeks of SNI with a bulb syringe, SNI with a nasal irrigation pot, and a control group of reflexology massage. Hypertonic saline was used in both treatment groups. Subjective questionnaires were administered at baseline and at the end of the study period. Both groups significantly improved, with no significant difference between the two SNI devices. Patients equally preferred the two devices.

Popular HVSI and LVSI formulations with patients and physicians are NeilMed® Sinus Rinse™ and Salinex®, respectively. These are two examples of positive pressure treatments, which have enjoyed widespread usage in North America preceding sufficient evidence-based medicine demonstrating safety and efficacy. This is likely because topical saline sprays are considered safe; they do not require a prescription and perhaps most importantly the massive marketing campaign surrounding SNI devices. SNI devices have received significant news coverage and appearances on major television shows, including the Oprah Winfrey Show, the New York Times, and numerous internet videos.

PURPOSE: The purpose of this study is to determine if there is a clinical benefit of high volume saline nasal irrigation (HVSI) over low volume saline irrigation (LVSI) in the postoperative period in patients with chronic Rhinosinusitis (CRS). This study is part of a multicenter collaborative project initiated by Macdonald et al. However, the sample size was not considered sufficient to conclude any significantly different effect between the two saline volumes (i.e. 86 participants); it was determined that a sample size of 176 (88 in each condition) was required (see attached in Section 9.8). To achieve this, our role is to collect data (plus those of four other Canadian rhinology research centres) from 20 patients and add our findings to theirs to establish an acceptable and significant result. This information would help otolaryngologists, family physicians, and other health care professionals recommend the best post-operative SNI (saline nasal irrigation) device for their patients with CRS.

HYPOTHESES: We hypothesize that there is an advantage of HVSI (NeilMed® Sinus Rinse™) over LVSI (Salinex®) in the early post-operative management in patients with chronic rhinosinusitis. The mechanical effect of high volume irrigation helps ensure that a larger surface area of sinonasal mucosa is debrided and cleansed.

RESEARCH METHOD: This is a multicenter, randomized, single blind, controlled prospective study evaluating the subjective and objective outcomes of HSVI versus LSVI in patients who have endoscopic sinus surgery (ESS) for CRS. One month postoperative scores will be compared to preoperative scores. The expected total number of patients to be enrolled in this study is approximately 100 (20 patient per 5 institutions), with a planned completion time of one year. We will approach 20 patients who are offered ESS for CRS for our part of the study.

Pre-operative documents will include a consent form to participate in the research study, two subjective questionnaires (SNOT-22 and Nasal and Sinus Symptom Score) to be completed by the patient and an objective endoscopy scale (POSE) to be completed by the surgeon. Preoperative CT scans are usually obtained in patients having ESS for CRS. These will be graded using the Lund-McKay score. Finally, endoscopic sinonasal photos will be taken if resources at the specific institution allow it. These scales are described in further detail below.

Evaluation Tests The Sinonasal Outcome Test-22 (SNOT-22) survey is a rhinology-specific quality of life instrument, based on 22 items. It is a subjective scale that is completed by the patient. A lower score represents a better quality of life. The SNOT-22 is commonly used in clinical research, and is reliable, valid, responsive, and easy to use.

The Nasal and Sinus Symptom Score is a rhinology-specific questionnaire based on 5 items. Patients rate the severity of these symptoms from "None" to "Severe".

The Perioperative Sinus Endoscopy (POSE) scoring system was developed in Canada and is used to endoscopically assess the sinonasal cavities of patients who have had ESS. The surgeon assesses the inflammatory status of the sinonasal cavity contents, including the middle turbinate, the middle meatus, ethmoid cavity, frontal recess/sinus and sphenoid sinus. Each site is graded from 0 to 2 depending on the degree of inflammation and/or purulence seen. A total score is calculated out of a total of up to 20, depending on the extent of surgery. This scale has compared well with other similar validated scales such as the Lund-McKay endoscopy staging system.

The Lund-McKay score is used to quantify sinonasal inflammation on a CT scan. Each of the following is given a score of 0-2 depending on the degree of opacification: anterior ethmoids, posterior ethmoids, maxillary sinus, sphenoid sinus, frontal sinus, and osteomeatal unit. At total score is calculated out of 24, a high score indicating more severe disease. This scale is also widely used in the assessment of CRS, and is reliable and valid.

Intervention/Treatment:

On the day of the surgery, patients will be provided with a box containing either a HVSI (NeilMed SINUS RINSE) or LVSI (Salinex®). The patient will be randomized using a computer software program, and the box containing the spray will be the same regardless of which one is used. The directions will be the same irrespective of the system given: two sprays in each nostril two times daily.

In this way the surgeon will be blinded to whether the patient has a HVSI or LVSI. The patient will be clearly instructed to NOT tell the surgeon which device they were given. In addition, surgeons involved in the study will be instructed to NEVER ask the patient which device they used.

Harms and discomforts:

Saline irrigation, HVSI or LVSI, is considered a safe treatment with no adverse effects. Occasionally patients will feel some discomfort, but it is a well-tolerated therapy. We do not perceive any risks with this treatment.

Patients may withdraw from the study at any time for any reason. This will not affect patient care in any way.

Sinus surgeons routinely prescribe medications in the preoperative period, including antibiotics and topical and/or systemic steroids. Surgeons will be instructed to treat their patients, preoperatively as they normally would, with no alteration in treatment other than the randomized saline irrigation bottle.

At one month postoperatively, patients will be reassessed in the clinic. The SNOT-22, Nasal and Sinus Symptoms Score (by patients), and POSE (by surgeons) questionnaires will be completed, and endoscopic photos will be taken.

Preoperative and one-month postoperative SNOT-22, Nasal and Sinus Symptoms Score, and POSE scores for the HVSI and LVSI will be compared to determine if there is a significant difference in subjective and/or objective outcomes. Patients will be stratified according to disease severity using the preoperative questionnaires and the Lund-McKay score to determine if patients with varying disease severity benefit more from one delivery device over the other.

We hope to involve 5 sinus surgeons across Canada, mostly from academic tertiary care institutions. Each surgeon will involve 20 patients in this study, for a total study recruitment of 100 patients. Each surgeon will submit a proposal to his/her own institution's Research Ethics Board.

The data from all 5 surgeons will be collected by the primary investigator (AJ). Data will be sent in a confidential manner over secure fax. Patient names and other specific identifiers will not be included with correspondence.

PROPOSED DATA ANALYSIS: Data will be entered into an Excel spreadsheet and statistical analysis will be applied with the Statistical Package for the Social Sciences (SPSS) vs.13. A total sample size was calculated at 100 patients (5 surgeons, 20 patients per surgeon at each institution) that would yield a useful and achievable analysis without being overly cumbersome. Because of the lack of research in this area, to achieve these study numbers alone would represent a significant achievement. Subsequently, data from these 100 patients would be added to those of the previously determined 86 (which will be sent by Dr. Macdonald in Toronto), placed onto the same spreadsheet and analyzed.

Implications of research: As stated above, our results may provide needed evidence for a common trend among Otolaryngologists. This will be the first study to document the value of different volume spray to treat postoperative sinus surgery; the results are potentially publishable in a major journal and would represent a major collaborative effort among Canadian Otolaryngologists. It would help maintain the University of British Columbia's and the Division of Otolaryngology's reputation in world-class research.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of unilateral or bilateral CRS
* Documented failed medical treatment of CRS
* 18 to 65 years of age
* Planned ESS for the treatment of CRS
* Able to read and understand English

Exclusion Criteria:

* Pregnant
* Cystic Fibrosis
* Diagnosed immotile cilia syndrome
* Diagnosed immunodeficiency syndrome
* Diagnosed fungal sinusitis
* Sinonasal tumours or obstructive lesions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change of preoperative from postoperative CT endoscopic photo scans used to evaluate different saline irrigation treatment volumes in patients with chronic rhinosinusitis. | 30 min at enrollment and 20 minutes at 1-month postoperative follow-up
  The value of either the HVSI or the LVSI to improve recovery and treatment of CRS postoperatively will be assessed.
Change of preoperative from postoperative sinus surgery regarding quality of life based on SNOT-22 questionnaire. | 15 min at enrollment and 10 minutes at 1-month postoperative follow-up
  A standard questionnaire, SNOT-22, will document improvements regarding quality of life.
Change of preoperative from postoperative sinus surgery regarding quality of life based on the Nasal and Sinus Symptoms Score questionnaire. | 15 min at enrollment and 10 minutes at 1-month postoperative follow-up
  A standard questionnaire, Nasal and Sinus Symptoms Score, will document improvements regarding quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Janjua, MD, Principal Investigator — Vancouver Coastal Health
Locations (1):
- Vancouver General Hospital/Otolaryngology Clinic, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Chen Y, Dales R, Lin M. The epidemiology of chronic rhinosinusitis in Canadians. Laryngoscope. 2003 Jul;113(7):1199-205. doi: 10.1097/00005537-200307000-00016. PMID 12838019
- [Background] Anand VK. Epidemiology and economic impact of rhinosinusitis. Ann Otol Rhinol Laryngol Suppl. 2004 May;193:3-5. doi: 10.1177/00034894041130s502. PMID 15174752
- [Background] Ray NF, Baraniuk JN, Thamer M, Rinehart CS, Gergen PJ, Kaliner M, Josephs S, Pung YH. Healthcare expenditures for sinusitis in 1996: contributions of asthma, rhinitis, and other airway disorders. J Allergy Clin Immunol. 1999 Mar;103(3 Pt 1):408-14. doi: 10.1016/s0091-6749(99)70464-1. PMID 10069873
- [Background] Van Cauwenberge P, Watelet JB. Epidemiology of chronic rhinosinusitis. Thorax. 2000 Oct;55 Suppl 2(Suppl 2):S20-1. doi: 10.1136/thorax.55.suppl_2.s20. No abstract available. PMID 10992549
- [Background] Tomooka LT, Murphy C, Davidson TM. Clinical study and literature review of nasal irrigation. Laryngoscope. 2000 Jul;110(7):1189-93. doi: 10.1097/00005537-200007000-00023. PMID 10892694
- [Background] Rabago D, Zgierska A, Mundt M, Barrett B, Bobula J, Maberry R. Efficacy of daily hypertonic saline nasal irrigation among patients with sinusitis: a randomized controlled trial. J Fam Pract. 2002 Dec;51(12):1049-55. PMID 12540331
- [Background] Meltzer EO, Hamilos DL. Rhinosinusitis diagnosis and management for the clinician: a synopsis of recent consensus guidelines. Mayo Clin Proc. 2011 May;86(5):427-43. doi: 10.4065/mcp.2010.0392. Epub 2011 Apr 13. PMID 21490181
- [Background] Lavigne F, Alizadehfar R, Balter Met al. Optimizing the usage of saline nasal irrigation (SNI) in the management of common respiratory conditions: from clinical evidence to daily practice. Unpublished, submission in progress 2011.
- [Background] Krayenbuhl M, Seppey M. [Efficacy of Rhinomer Force 3 in the postoperative course of endonasal surgery]. Rev Med Suisse Romande. 1995 Mar;115(3):249-52. No abstract available. French. PMID 7777766
- [Background] Seppey M, Schweri T, Hausler R. Comparative randomised clinical study of tolerability and efficacy of Rhinomer Force 3 versus a reference product in post-operative care of the nasal fossae after endonasal surgery. ORL J Otorhinolaryngol Relat Spec. 1996 Mar-Apr;58(2):87-92. doi: 10.1159/000276805. PMID 8736053
- [Background] Pigret D, Jankowski R. Management of post-ethmoidectomy crust formation: randomized single-blind clinical trial comparing pressurized seawater versus antiseptic/mucolytic saline. Rhinology. 1996 Mar;34(1):38-40. PMID 8739868
- [Background] Harvey RJ, Debnath N, Srubiski A, Bleier B, Schlosser RJ. Fluid residuals and drug exposure in nasal irrigation. Otolaryngol Head Neck Surg. 2009 Dec;141(6):757-61. doi: 10.1016/j.otohns.2009.09.006. PMID 19932850
- [Background] Harvey RJ, Goddard JC, Wise SK, Schlosser RJ. Effects of endoscopic sinus surgery and delivery device on cadaver sinus irrigation. Otolaryngol Head Neck Surg. 2008 Jul;139(1):137-42. doi: 10.1016/j.otohns.2008.04.020. PMID 18585576
- [Background] Heatley DG, McConnell KE, Kille TL, Leverson GE. Nasal irrigation for the alleviation of sinonasal symptoms. Otolaryngol Head Neck Surg. 2001 Jul;125(1):44-8. doi: 10.1067/mhn.2001.115909. PMID 11458213
- [Background] Sweeney C. Short, Stout, Has a Handle on Colds. Available at: http://www.nytimes.com/2008/01/03/fashion/03skin.html. Accessed September 5th, 2011. Published Jan. 3rd, 2008.
- [Background] Morley AD, Sharp HR. A review of sinonasal outcome scoring systems - which is best? Clin Otolaryngol. 2006 Apr;31(2):103-9. doi: 10.1111/j.1749-4486.2006.01155.x. PMID 16620328
- [Background] Wright ED, Agrawal S. Impact of perioperative systemic steroids on surgical outcomes in patients with chronic rhinosinusitis with polyposis: evaluation with the novel Perioperative Sinus Endoscopy (POSE) scoring system. Laryngoscope. 2007 Nov;117(11 Pt 2 Suppl 115):1-28. doi: 10.1097/MLG.0b013e31814842f8. PMID 18075447
- [Background] Hopkins C, Browne JP, Slack R, Lund V, Brown P. The Lund-Mackay staging system for chronic rhinosinusitis: how is it used and what does it predict? Otolaryngol Head Neck Surg. 2007 Oct;137(4):555-61. doi: 10.1016/j.otohns.2007.02.004. PMID 17903570
- [Background] Desrosiers M, Evans GA, Keith PK, Wright ED, Kaplan A, Bouchard J, Ciavarella A, Doyle PW, Javer AR, Leith ES, Mukherji A, Robert Schellenberg R, Small P, Witterick IJ. Canadian clinical practice guidelines for acute and chronic rhinosinusitis. J Otolaryngol Head Neck Surg. 2011 May;40 Suppl 2:S99-193. English, French. PMID 21658337
- [Result] Macdonald KI, Wright ED, Sowerby LJ, Rotenberg BW, Chin CJ, Rudmik L, Sommer DD, Nayan S, DesRosiers M, Tewfik MA, Valdes CJ, Massoud E, Thomas D, Kilty SJ, Vescan A, Mechor B, Lavigne F, Fandino M, Javer AR, Witterick IJ. Squeeze bottle versus saline spray after endoscopic sinus surgery for chronic rhinosinusitis: a pilot multicentre trial. Am J Rhinol Allergy. 2015 Jan-Feb;29(1):e13-7. doi: 10.2500/ajra.2015.29.4125. PMID 25590308